CLINICAL TRIAL: NCT03323528
Title: A Multi-centre, Randomized, Placebo-controlled, Double-blind, Parallel-group Study Investigating Safety and Efficacy of a Sore Throat Lozenge in the Symptomatic Treatment of Patients With Acute Pharyngitis
Brief Title: Safety and Efficacy of a Sore Throat Lozenge DORITHRICIN in Patients With Acute Pharyngitis
Acronym: DoriPha
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Collaborators: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-003962-24
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-10

CONDITIONS: Pharyngitis
Keywords: Dorithricin; Tyrothricin; Benzalkonium chloride; Benzocaine; placebo-controlled; Pharyngitis; sore throat; throat pain; difficulty swallowing; complete responder; lozenge; Non-streptococcal Infections
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: randomized allocation of participants to verum or placebo (1:1)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: investigation: participant, care provider and investigator blinded assessment: participant, care provider and investigator blinded outcome analysis: statistician blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dorithricin (Active Comparator): Dorithricin throat lozenges is a fixed combination of three active substances: Benzalkonium Chloride-Benzocaine Topical plus tyrothricin. Lozenge has to be sucked slowly until it fully dissolves in the mouth and dosed up to 8 lozenges per day. Test product without mint oil.
  Intervention: The initial dose is administered at the study site. Patients administer at home 1 lozenge at intervals of 2 hours (±15 minutes) up to a maximum of 8 lozenges per day.
  Interventions: Drug: Benzalkonium Chloride-Benzocaine Topical
- Placebo (Placebo Comparator): Placebo Oral Tablet is taken orally. Placebo consists of a lozenge with matched appearance and the same excipients as those of the Dorithricin lozenge. The initial dose (2 lozenges simultaneously) is administered at the study site.
  Intervention: Patients are instructed to administer at home 1 lozenge at intervals of 2 hours (±15 minutes) up to a maximum of 8 lozenges per day.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Benzalkonium Chloride-Benzocaine Topical — Dorithricin = tyrothricin, benzalkonium chloride, benzocaine
  Other Names: triple combination
  Arms: Dorithricin
Drug: Placebo Oral Tablet — Placebo Oral Tablet = a lozenge with matched appearance and the same excipients as Active Comparator Dorithricin lozenge.
  Intervention: Patients are instructed to administer at home 1 lozenge at intervals of 2 hours (±15 minutes) up to a maximum of 8 lozenges per day.
  Other Names: Placebo lozenge
  Arms: Placebo

SUMMARY:
The aim of this multi-center, randomized, double-blind, placebo-controlled trial is to compare the efficacy and safety of Dorithricin® lozenge - a triple combination of 0.5 mg tyrothricin, 1.0 mg benzalkonium chloride, and 1.5 mg benzocaine - in repeat dosing for 3 days to matched placebo lozenges in the treatment of acute pharyngitis in adults.

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled trial, adult patients with non-streptococcal sore throat and signs of moderate-to-severe associated pain (pain intensity on the 11-point Sore Throat Pain Intensity Scale NRS ≥7 and ≥50 mm on the subjective 0-100 mm visual analogue) are assigned to Dorithricin® or matching placebo lozenge treatment. Efficacy was assessed at the investigating center for 2 hrs after first dosing, and 3 days later (visit 2). The primary efficacy end-point is the percentage of total responders assessed at visit 2, i.e. complete resolution of throat pain and difficulty in swallowing at approx. 72 hrs after first application of treatment, Safety and local tolerability are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients aged ≥18 years
* Signed informed consent form
* Clinically diagnosed acute pharyngitis (TPA ≥5)
* Recent onset of symptoms (≤24 hours)
* Pain intensity of ≥8 on an 11-point NRS
* Difficulty in swallowing (100-mm VAS ≥50 mm)

Exclusion Criteria:

* Patients with strong suspicion of streptococcus A infection (McIsaac score ≥3)
* Positive rapid streptococcus A test (rapid antigen detection test) to exclude the major bacterial pathogen responsible for sore throat
* Purulent tonsillitis
* The use of systemic/local antibiotics in the throat area within 7 days prior to screening and during the study
* The use of any systemic analgesics/local analgesics in the throat area (e.g. non-steroidal drugs, [acetylsalicylic acid >100 mg], paracetamol) within 36 hours prior to screening and during the study
* The use of local anaesthetics for treatment of sore throat within 2 days prior to screening and during the study
* The use of any systemic anti-inflammatory drug/local anti-inflammatory drug in the throat area (e.g. glucocorticoids) within 4 weeks prior to screening and during the study
* The use of any other 'sore throat medication' (e.g., lozenges, drops, sprays) or other 'cold medication' that could have interfered with the results of the study within 7 days prior to screening and during the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
percentage of total responders assessed at Visit 2 (72 hours after first treatment) | 72 hours after first treatment
  complete resolution of throat pain and difficulty in swallowing at Visit 2

SECONDARY OUTCOMES:
percentage of total responders assessed after 48 hours after first treatment | 48 hours after first treatment
  complete resolution of throat pain and difficulty in swallowing after 48 hours after first treatment
percentage of patients with complete resolution of throat pain 72 hours after first treatment | 72 hours after first treatment
  complete resolution of throat pain after 72 hours after first treatment
percentage of patients with complete resolution of difficulty in swallowing 72 hours after first treatment | 72 hours after first treatment
  complete resolution of difficulty in swallowing after 72 hours after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: R Ammer, MD, PhD, Study Director — MEDICE Arzneimittel Puetter GmbH&Co.KG; R Ammer, MD, PhD, Study Director — Universtiy hospital Muenster, MedD
Locations (1):
- doc-HNO for the DoriPha investigators, Röthenbach an der Pegnitz, Germany

IPD SHARING:
Plan to Share IPD: No
study protocol, statistical analysis plan, informed consent form, clinical study report are shared with all 26 recruited centers of the DoriPha investigators

REFERENCES:
- [Derived] Palm J, Fuchs K, Stammer H, Schumacher-Stimpfl A, Milde J; DoriPha investigators. Efficacy and safety of a triple active sore throat lozenge in the treatment of patients with acute pharyngitis: Results of a multi-centre, randomised, placebo-controlled, double-blind, parallel-group trial (DoriPha). Int J Clin Pract. 2018 Dec;72(12):e13272. doi: 10.1111/ijcp.13272. Epub 2018 Oct 17. PMID 30329199
- See also: Test product description — http://www.dorithricin.de